CLINICAL TRIAL: NCT00635063
Title: A Multicentre, Randomised, Double-Blind, Double-Dummy, Crossover Study to Evaluate the Safety and Efficacy of AD 923 (Fentanyl Sublingual) in Comparison to Morphine Sulphate Immediate Release (MSIR) for the Treatment of Breakthrough Pain in Subjects With Malignancies
Brief Title: A Multicentre Study to Evaluate the Safety and Efficacy of AD 923 in Comparison to MSIR for the Treatment of CBP in Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination is due to a combination of a device defect potentially impacting the quality of the AD 923 IMP and a major change in corporate strategy.
Sponsor: Sosei (Industry)
Responsible Party: Dr Robin Bannister, Sosei R&D Ltd
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-AD923-005
Record Dates: First submitted 2008-03-04; First posted 2008-03-13 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Cancer; Pain
Keywords: Cancer Breakthrough Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AD 923 (Experimental)
  Interventions: Drug: AD 923
- MSIR (Active Comparator)
  Interventions: Drug: AD 923

INTERVENTIONS:
Drug: AD 923

SUMMARY:
Purpose:

The purpose of this study is to compare the efficacy and safety of AD 923 to the most widely used current treatment (MSIR) in the management of target BTP in subjects with malignancies who are taking a stable dose of background opioids. The efficacy evaluation criteria have been designed to determine whether AD 923 provides superior analgesia compared with MSIR as measured by the primary endpoint.

ELIGIBILITY:
Main Inclusion Criteria:

* The subject is a male or female, at least 18 years of age.
* The subject has a malignancy, is receiving opioid therapy for his or her underlying persistent cancer pain, and is tolerant to the opioid therapy.
* The subject typically has 2 to 6 episodes of target BTP per day that require treatment.
* The subject has a life expectancy of >3 months.
* The subject or his or her caregiver has easy, reliable access to a telephone.

Main Exclusion Criteria:

* The subject is a female who is pregnant or lactating.
* The subject has any respiratory or cardiac condition that, in the opinion of the investigator, may be clinically worsened by opioids.
* The subject has any allergy to the AD 923 product or excipients, namely: fentanyl, dehydrated alcohol, menthol, saccharin, and citrate buffer; or to the MSIR product excipients, namely: morphine sulphate, lactose (anhydrous), pregelatinized maize starch, povidone, purified water, magnesium stearate, talc, and tablet coatings.
* The subject has any neurological or psychiatric disease that, in the opinion of the investigator, would compromise data collection.
* The subject has uncontrolled or rapidly escalating pain.
* The subject has any significant laboratory test results that, in the opinion of the investigator, will compromise subject safety or the conduct of the study.
* The subject has plans to undergo chemotherapy, radiotherapy, or surgery during the treatment period. The exception is that subjects may continue chemotherapy over the study period, provided it is not expected to alter the pain state or response to pain medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
To evaluate the efficacy of AD 923 in comparison to MSIR in the management of breakthrough pain in subjects with malignancies who are taking a stable dose of background opioids.

SECONDARY OUTCOMES:
To assess the safety and tolerability of AD 923 in the management of breakthrough pain in subjects with malignancies who are taking a stable dose of background opioids.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MBBS, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Sosei R&D Ltd, Saffron Walden, Essex, United Kingdom